CLINICAL TRIAL: NCT02593240
Title: Worksite Wellness Study
Brief Title: Worksite Wellness Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Sai Krupa Das, Scientist, Tufts University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 11768
Record Dates: First submitted 2015-10-21; First posted 2015-11-02 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Obesity; Overweight; Quality of Life
Keywords: Energy; Presenteeism; Absenteeism; Cardiometabolic health; Obesity; Overweight; Weight Loss; Quality of Life; Weight Control; Eating Behavior; Food Cravings; Hunger; Worksite Wellness
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Human Performance Institute© (Experimental): These participants will be part of the intervention sites and will receive the Human Performance Institute© intervention for the duration of the study (18 months).
  Interventions: Behavioral: Human Performance Institute©
- The iDiet® with Voucher (Experimental): These participants will be part of the intervention sites and will receive the iDiet® with Voucher for the duration of the study (18 months).
  Interventions: Behavioral: The iDiet® (also called Healthy Weight for Living when used as a not-for-profit intervention) with Voucher
- The iDiet® with Food (Experimental): These participants will be part of the intervention sites and will receive the iDiet® with Food for the duration of the study (18 months).
  Interventions: Behavioral: The iDiet® (also called Healthy Weight for Living when used as a not-for-profit intervention) with Food
- Wait-listed control (No Intervention): These participants will be part of the control sites and will participate in outcome assessments for a 6-month period only.

INTERVENTIONS:
Behavioral: The iDiet® (also called Healthy Weight for Living when used as a not-for-profit intervention) with Food — The intensive iDiet® group behavioral weight loss program will be delivered in person at the worksite or by videoconference and with support of the program's web platform. This intervention will be delivered by trained group leaders and will initially include weekly 1-hour support and education meetings of 20 participants/group with a message board for group communication and individual communication with the group leader. Over time support will be provided online rather than in live meetings. The intervention involves a weight loss behavioral program with particular emphasis on hunger reduction and craving control for both weight loss and prevention of weight regain. Half of the participants per worksite receiving the iDiet® intervention will be randomized to receive commercial dried food products (partial supply) from Yevo Intl., which are designed to help with weight control and health.
  Arms: The iDiet® with Food
Behavioral: The iDiet® (also called Healthy Weight for Living when used as a not-for-profit intervention) with Voucher — The intensive iDiet® group behavioral weight loss program delivered in person at the worksite or by videoconference and with support of the program's web platform. This intervention will be delivered by trained group leaders and will initially include weekly 1-hour support and education meetings of 20 participants/group with a message board for group communication and individual communication with the group leader. Over time support will be provided online rather than in live meetings. The intervention involves a weight loss behavioral program with particular emphasis on hunger reduction and craving control for both weight loss and prevention of weight regain. Half of the participants per worksite receiving the Diet® intervention will be randomized to receive gift cards monthly for the first 6 months to purchase foods at their local grocery store (partial costs).
  Arms: The iDiet® with Voucher
Behavioral: Human Performance Institute© — The Human Performance Institute© (HPI) training workshop is a comprehensive individual development training program that focuses on the concept of energy management. The primary aim of this program is to help individuals develop attitudes, habits, and behaviors that increase their levels of daily energy, life satisfaction, and overall functioning. The course is delivered at an off-site location over 2.5 days, by 3 coaches, in a group format of 25 - 32 participants (with employees from more than one worksite per group).
  Arms: Human Performance Institute©

SUMMARY:
Worksites offer attractive locations for reducing the national prevalence of overweight and obesity. Interventions that are both effective and sustainable for producing long-term changes in health and employee wellness are urgently needed. In an 18-month worksite randomized controlled trial in 12 worksites, this study will test two lifestyle approaches designed to facilitate behavior modification for achieving long-term improvements in health and quality of life. Worksites randomized to the immediate intervention arm will receive the two on-site wellness programs and the randomized control sites will participate in outcomes assessments for the initial 6-month period, after which participants will receive vouchers to participate in the program of their choice. The primary focus of the worksite wellness study is to identify ways to improve health-related quality of life, with a particular focus on a decrease in cardiometabolic risk factors, including weight, improved weight-related wellness, and improved energy level in work and life. The two interventions will be separately tested against the control condition in intention-to-treat models and with a completers analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to sign an informed consent form
2. Willingness to provide release from his/her physician before starting the intervention program-a requirement for each of the 3 wellness programs
3. Willingness to provide email identification (ID) and contact information to the commercial program facilitators to receive program materials and other feedback related to program progress
4. Willingness to complete outcome assessments and self-monitoring in order to track intervention effectiveness
5. BMI ≥ 20 kg/m2 and < 50 kg/m2 at screening, if participant opts into the HPI arm
6. BMI ≥ 25 kg/m2 and < 50 kg/m2 at screening, if participant opts into the weight loss arm

Exclusion Criteria:

1. Employees who are temporary contract workers or employees who work remotely most of the time
2. < 21 years of age
3. Participation in a weight loss program or intensive wellbeing program at time of enrollment
4. Pregnant or lactating (per self-reports, now or intended during study)
5. Prior weight loss surgery or a medical complication that would prevent full participation
6. Multiple severe dietary intolerances (e.g. gluten combined with dairy or meat) which would reduce intervention adherence
7. Non-English speaking
8. Individuals who have lost > 15 pounds in the past 6 months
9. Mobility limitations (inhibiting the ability to stand on one's own or get on and off of the scale)
10. Major diseases including active cancer or cardiovascular disease
11. BMI < 25 kg/m2 or ≥ 50 kg/m2 at screening, for those that opt-in to the weight-loss group
12. BMI <20 kg/m2 or ≥ 50 kg/m2 at screening, for those that opt-in to the HPI group

    For those interested in the weight loss intervention, additional exclusion criteria are as follows:
13. Any condition that influences the ability to absorb food (e.g. inflammatory bowel disease or celiac disease)
14. Very active individuals (> 2 hours/day or >14 hours/week of vigorous activity).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Weight (iDiet/Healthy Weight for Living arms) | 1.5 years
  Fasted measurements of weight obtained in duplicate to ±0.1 kg at baseline, 6, 12, and 18 months using the TANITA TBF-300A.
Quality of Life (HPI arm) | 1.5 years
  Assessed by the RAND Short Form 36 Health Survey (SF-36) at baseline, 6, 12, and 18 months.

SECONDARY OUTCOMES:
Blood pressure | 1.5 years
  Systolic and diastolic blood pressure (mm Hg) measured to the nearest 1 mm Hg at baseline, 6, 12, and 18 months using a validated automated monitor (3 fasted measurements, 5 minutes apart, after 5 minutes of quiet sitting).
Cholesterol | 1.5 years
  Total cholesterol, high-density lipoprotein, and low-density lipoprotein measured at baseline, 6, 12, and 18 months using the Alere Cholestech LDX® System, which requires 40 microliters of blood (fasted lipid panel).
Triglycerides | 1.5 years
  Triglycerides measured at baseline, 6, 12, and 18 months using the Alere Cholestech LDX® System (fasted lipid panel).
Glucose | 1.5 years
  Fasting blood glucose measured at baseline, 6, 12, and 18 months using the Alere Cholestech LDX® System.
Hemoglobin A1c | 1.5 years
  HbA1c measured at baseline, 6, 12, and 18 months using the Siemens DCA Vantage, which requires 1 microliter of blood (fasted measurement).
Eating behavior (Food Preferences) | 1.5 years
  Assessed by the Food Preferences Questionnaire (self-administered) at baseline, 6, 12, and 18 months.
Eating behavior (Three-Factor Eating) | 1.5 years
  Assessed by the Three-Factor Eating Questionnaire (self-administered) at baseline, 6, 12, and 18 months.
Eating behavior (Food Cravings) | 1.5 years
  Assessed by the Food Cravings Questionnaire - Trait (self-administered) at baseline, 6, 12, and 18 months.
Depression | 1.5 years
  Assessed by the Center for Epidemiological Studies Depression Scale (self-administered) at baseline, 6, 12, and 18 months.
Mood | 1.5 years
  Assessed by the Profile of Mood States (self-administered) at baseline, 6, 12, and 18 months. Variables include anger-hostility, depression-dejection, fatigue-inertia, and vigor-activity.
Physical Activity | 1.5 years
  Assessed by the International Physical Activity Questionnaire (self-administered) at baseline, 6, 12, and 18 months.
Well-being | 1.5 years
  Assessed by the Ryff Purpose in Life scale (self-administered) at baseline, 6, 12, and 18 months.
Productivity | 1.5 years
  Assessed by the Work Productivity and Impairment scale (self-administered) at baseline, 6, 12, and 18 months.
Sleep | 1.5 years
  Assessed by the Medical Outcomes Study Sleep Questionnaire (self-administered) at baseline, 6, 12, and 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Krupa Das, PhD, Principal Investigator — Tufts University; Susan B Roberts, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University Human Nutrition Research Center on Aging, Boston, Massachusetts, United States